CLINICAL TRIAL: NCT02788552
Title: Optimum Thiamine Intervention (OpT In) for Treatment and Prevention of Wernicke-Korsakoff Syndrome (WKS): A Randomised Controlled Trial
Brief Title: Optimum Thiamine Intervention (OpTIn) Trial
Acronym: OpTIn
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-08-27_Version2.1; ACTRN12614000327684 (Registry Identifier: ANZCTR); Project Grant GNT1057968 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2014-09-26; First posted 2016-06-02 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Wernicke-Korsakoff Syndrome
Keywords: Neurological; Diet and Nutrition; Mental Health
MeSH Terms: conditions — Korsakoff Syndrome; Neurologic Manifestations; Psychological Well-Being | interventions — thiamine hydrochloride; Thiamine; Vitamin B Complex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Acute Symptomatic WKS- 300mg (Active Comparator): Thiamine Hydrochloride 300mg daily (i.e. 100mg 3 times/day) for 5 days
  Interventions: Drug: Thiamine Hydrochloride
- Acute Symptomatic WKS - 900mg (Active Comparator): Thiamine Hydrochloride 900mg daily (i.e. 300mg 3 times/day) for 5 days
  Interventions: Drug: Thiamine Hydrochloride
- Acute Symptomatic WKS - 1500mg (Active Comparator): Thiamine Hydrochloride 1500mg daily (i.e. 500mg 3 times/day) for 5 days.
  Interventions: Drug: Thiamine Hydrochloride
- High-risk subclinical WKS- 100mg (Active Comparator): Thiamine Hydrochloride 100mg once daily for 3 days.
  Interventions: Drug: Thiamine Hydrochloride
- High-risk subclinical WKS- 300mg (Active Comparator): Thiamine Hydrochloride 300mg (i.e. 100mg 3 time/day) for 3 days
  Interventions: Drug: Thiamine Hydrochloride
- High-risk subclinical WKS - 900mg (Active Comparator): Thiamine Hydrochloride 900mg daily (i.e. 300mg 3 times/day) for 3 days.
  Interventions: Drug: Thiamine Hydrochloride

INTERVENTIONS:
Drug: Thiamine Hydrochloride — Administered Intravenously in 100ml bag of normal saline (0.9%) infused over 30 mins.
  Other Names: Vitamin B1; Thiamine Chloride; Aneurine Hydrochloride; B Complex Vitamin

SUMMARY:
Wernicke-Korsakoff syndrome (WKS), once thought to be a rare condition, is now known to be common in people with nutritional deficiencies or alcohol dependence. The primary cause of WKS is thiamine deficiency, and more than 90% of cases are reported in alcohol dependent patients because alcohol dependence predisposes to severe nutritional deficiency. WKS may lead to significant, long-term brain dysfunction with severe effects on work, personal and social function. Whilst effective treatment may greatly reduce severe disability and the human and social costs of this illness, almost no evidence exists on optimal dosing regimens. This project proposes to develop quality evidence for effective treatment of WKS in an Aboriginal setting.

DETAILED DESCRIPTION:
Wernicke-Korsakoff syndrome (WKS), once thought to be a rare condition, is now known to be common in people with nutritional deficiencies or alcohol dependence. The primary cause of WKS is thiamine deficiency, and more than 90% of cases are reported in alcohol dependent patients because alcohol dependence predisposes to severe nutritional deficiency. WKS may lead to significant, long-term brain dysfunction with severe effects on work, personal and social function. Whilst effective treatment may greatly reduce severe disability and the human and social costs of this illness, almost no evidence exists on optimal dosing regimens. This project proposes to develop quality evidence for effective treatment of WKS in an Aboriginal setting..

The need for evidence-based thiamine treatment protocols is of great clinical importance for two related reasons. First, in relation to acute symptomatic WKS, a failure to treat immediately or adequately may result in profound and often permanent cognitive and neurological disability. Secondly, the need for evidence-based treatment guidelines is greatly magnified when it is recognised that milder, subclinical WKS may be preventable with adequate thiamine treatment.

The aims of this study are to determine the optimal thiamine dose required for:

A. Treatment of acute symptomatic WKS among Aboriginal and non-Aboriginal alcohol dependent patients.

B. Reducing or preventing subclinical WKS-related brain damage in at-risk Aboriginal and non-Aboriginal alcohol-dependent patients.

Primary Hypotheses

1. Among alcohol-dependent patients with acute symptomatic WKS, higher doses of parenteral thiamine (1500mg) will lead to greater improvements in specific cognition and neurological functions than lower doses (900mg or 300mg).
2. Among alcohol-dependent patients that are at high risk for subclinical WKS-related brain damage, higher doses of parenteral thiamine (900mg) will lead to greater improvements in specific cognition and neurological functions compared to lower doses (300mg or 100mg).

Secondary Hypotheses

1. Thiamine deficient patients will show poorer performance on cognitive and neurological measures.
2. Patients with concurrent magnesium deficiency will show greater impairment at baseline.
3. Nutritional risk and alcohol frequency will correlate with thiamine pyrophosphate levels.
4. Number of previous admissions with thiamine supplementation in the past 3 months will correlate with thiamine pyrophosphate levels

ELIGIBILITY:
Inclusion Criteria:

* Aged range 18-65 years
* History of heavy alcohol use AUDIT-C score >4 or consumption >60mg/day or >80mg/binge

Exclusion Criteria:

* Pregnant women
* Under the age of 18 or over 65 years old
* Known pre-existing neurological or cognitive impairment unrelated to thiamine deficiency or WKS
* Renal dialysis patients
* Sedated patients in ICU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2014-09; Primary Completion 2019-05-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Standardised Cognitive assessment - RUDAS | Days 1 and 5 for Acute symptomatic patients and Days 1 and 3 for at risk patients
  Evaluate differences in cognitive outcomes among acute symptomatic WKS patients under three parenteral thiamine treatment conditions (300mg/day for 5 days, versus 900mg/day for 5 days, versus 1500mg/day for 5 days); and among patients at high risk of subclinical WKS-related brain damage under three parenteral thiamine treatment conditions (100mg/day for 3 days, versus 300mg/day for 3 days, versus 900mg/day for 3 days); using Standardised cognitive assessment - Rowland Universal Dementia Assessment Scale (RUDAS).
Standardised Cognitive assessment - CogState | Days 1 and 5 for Acute symptomatic patients and Days 1 and 3 for at risk patients
  Evaluate differences in cognitive outcomes among acute symptomatic WKS patients under three parenteral thiamine treatment conditions (300mg/day for 5 days, versus 900mg/day for 5 days, versus 1500mg/day for 5 days); and among patients at high risk of subclinical WKS-related brain damage under three parenteral thiamine treatment conditions (100mg/day for 3 days, versus 300mg/day for 3 days, versus 900mg/day for 3 days); using CogState battery.
Standardised Cognitive assessment - Story Memory Recall Test | Days 1 and 5 for Acute symptomatic patients and Days 1 and 3 for at risk patients
  Evaluate differences in cognitive outcomes among acute symptomatic WKS patients under three parenteral thiamine treatment conditions (300mg/day for 5 days, versus 900mg/day for 5 days, versus 1500mg/day for 5 days); and among patients at high risk of subclinical WKS-related brain damage under three parenteral thiamine treatment conditions (100mg/day for 3 days, versus 300mg/day for 3 days, versus 900mg/day for 3 days); using Story Memory Recall test
Standardised neurological examination | Days 1 and 5 for acute symptomatic patients; Days 1 and 3 for at risk patients
  Evaluate differences in neurological outcomes among acute symptomatic WKS patients under three parenteral thiamine treatment conditions (300mg/day for 5 days, versus 900mg/day for 5 days, versus 1500mg/day for 5 days);and among patients at high-risk of subclinical WKS-related brain damage under three parenteral thiamine treatment conditions (100mg/day for 3 days, versus 300mg/day for 3 days, versus 900mg/day for 3 days); Using Standardised neurological examination. Aggregated as either normal or abnormal.

SECONDARY OUTCOMES:
Blood thiamine levels | Days 1 and 5 for acute symptomatic patients; days 1 and 3 for at risk patients
  Correlate changes in red cell thiamine test results (blood test) with cognitive (standardised cognitive assessments score) and neurological functioning (standardised neurological examination).
Magnesium levels | Days 1 and 5 for acute symptomatic patients; Days 1 and 3 for at risk patients
  Examine the impact of magnesium deficiency (magnesium blood test) on thiamine treatment response (cognition as measured by standardised cognitive assessments and thiamine pyrophosphate levels as measured by blood test).
Demographic factors | Day 1
  Assess independent predictors of WKS including nutritional factors, substance use history and demographic factors assessed by questionnaire items including Nutritional Risk Assessment and AUDIT-C.
Readmission | Day 1
  Examine the impact of patient re-admission on red cell thiamine pyrophosphate levels (blood test) and cognitive and neurological functioning (standardised cognitive and neurological assessments)

CONTACTS AND LOCATIONS:
Overall Officials: Kylie Dingwall, PhD, Principal Investigator — Menzies School of Health Research
Locations (1):
- Alice Springs Hospital, Alice Springs, Northern Territory, Australia

IPD SHARING:
Plan to Share IPD: No